CLINICAL TRIAL: NCT02832570
Title: Etude préliminaire Sur l'efficacité Aigue du Sildenafil Sur le Temps de Marche Chez Les Patients Atteints d'AOMI de Stade II présentant Une Claudication artérielle
Brief Title: Sildenafil Efficacy Study on Time Walk From Peripheral Arterial Desease Patients (Stade II) With Arterial Claudication
Acronym: ARTERIOFIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOI 2015-07
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2017-10

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sildenafil (Experimental): Single sildenafil oral intake (100 mg) approximately 2 hours before the treadmill test.
  Interventions: Drug: Sildenafil 100mg single oral dose
- Placebo (Placebo Comparator): Single placebo intake approximately 2 hours before the treadmill test.
  Interventions: Drug: Placebo, Oral intake single dose

INTERVENTIONS:
Drug: Sildenafil 100mg single oral dose — Measurement of maximal walking distance on a constant load treadmill test (3.12 km/ 10% slope)
  Other Names: Viagra verventi
  Arms: Sildenafil
Drug: Placebo, Oral intake single dose — Measurement of maximal walking distance on a constant load treadmill test (3.12 km/ 10% slope)
  Other Names: Sugar pills manufactured to mimick Sildenafil 100 mg
  Arms: Placebo

SUMMARY:
Efffect of a single dose oral intake of sildenafil Or placebo on the walking capacity on treadmill of PAD patients with claudication

DETAILED DESCRIPTION:
Sildenafil 100mg or Placebo Oral intake 2 hours before the treadmill test Safety and security control throughout the period of drug efficacy (approx 4 hours) Evaluation of maximal walking distance for a constant load treadmill test (3.2 kml/h 10% slope)

ELIGIBILITY:
Inclusion Criteria:

* Patient with peripheral arterial desease stade II
* Patient with vascular claudication for at least 3 months
* Patient able to perform a treadmill walking test with time to walk < 5min

Exclusion Criteria:

* Patient suffering from ischemia
* Previous angina or myocardial
* Patient treated with nitrates drugs
* Patient with severe renal insufficiency
* Patient with severe hepatic insufficiency
* Patient with hypotension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Walking duration on treadmill | 2 hours after treatment intake
  Treadmill test with consttant load procedure 3.2 km/h H 10% slope up to 15 minutes followed by incremental load according tpo the Bruce protocole thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Loukman OMARJEE, MD, Principal Investigator — University Hospital, Angers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omarjee L, Le Pabic E, Custaud MA, Fontaine C, Locher C, Renault A, Jaquinandi V, Azzola V, Barbeau-Terrier C, Laporte I, Ripoche M, Onillon Y, Chretien JM, Daniel V, Chao de la Barca JM, Homedan C, Reynier P, Abraham P, Mahe G. Effects of sildenafil on maximum walking time in patients with arterial claudication: The ARTERIOFIL study. Vascul Pharmacol. 2019 Jul-Aug;118-119:106563. doi: 10.1016/j.vph.2019.05.003. Epub 2019 May 30. PMID 31152977